CLINICAL TRIAL: NCT07105033
Title: Development and Pilot Trial of Focused ACT (FACT) for Patients With Advanced Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0481; NCI-2025-05620 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Examine Initial Acceptability and Efficacy Signal of FACT (Experimental): Potential participants will be identified weekly via MDACC's computerized appointment system for the Supportive Care Outpatient Clinic.
  Interventions: Behavioral: FACT Session
- Controlled Trial (RCT) to Examine Feasibility, Acceptability and Initially Efficacy of FACT (Experimental): Potential participants will be identified weekly via MDACC's computerized appointment system for the Supportive Care Outpatient Clinic.
  Interventions: Behavioral: Enhanced Usual Care and Assessments

INTERVENTIONS:
Behavioral: FACT Session — Participants will participate in 4 weekly, 35-45 minute sessions
  Arms: Examine Initial Acceptability and Efficacy Signal of FACT
Behavioral: Enhanced Usual Care and Assessments — Participants will complete a symptoms questionnaire
  Arms: Controlled Trial (RCT) to Examine Feasibility, Acceptability and Initially Efficacy of FACT

SUMMARY:
To learn about the effects of an intervention program called Focused Acceptance and Commitment Therapy (FACT) on the level of anxiety patients diagnosed with cancer feel about death.

To learn if an intervention program called Focused Acceptance and Commitment Therapy (FACT), designed to help reduce death-related anxiety, is effective and acceptable to patients diagnosed with advanced cancer.

DETAILED DESCRIPTION:
Primary Objectives:

Phase 1 To estimate the initial feasibility and acceptability of delivering the iteratively developed FACT in a single-arm pilot trial. We hypothesize that FACT will be both feasible (defined criteria: ≥90% on intervention fidelity ratings, attendance of ≥70% of FACT sessions, retention post-intervention assessment completion 70%) and acceptable (defined criteria: patients will report average satisfaction as ≥4/5; average appropriateness of the intervention as ≥4/5; ≥75% would recommend FACT to others, and ≥50% indicate they are likely to use FACT strategies following sessions).

Phase 2 To estimate initial within person change in self-report measures of death anxiety (DADDS) and cognitive fusion (CFQ) from baseline to post-treatment and 6-week follow-up assessment, in patients who participate in FACT intervention.

Secondary Objectives:

Phase 1 To estimate initial within person change in self-report measures of death anxiety (DADDS), death anxiety 2 item measure, cognitive fusion (CFQ), QOL (QUAL-E), anxiety (GAD-7), depression (CES-D), perceived stress (PSS), perceived social support (ISEL), illness understanding (Prigerson Illness Understanding Scale) and coping strategies (Brief COPE)) from baseline to post-treatment and 6-week follow-up assessment in patients who participate in FACT intervention in a single-arm pilot trial.

Phase 2 To estimate feasibility and acceptability of FACT in a pilot RCT. We hypothesize that FACT will be both feasible (defined criteria: ≥90% on intervention fidelity ratings, attendance of ≥70% of FACT sessions, retention post-intervention assessment completion 70%) and acceptable (defined criteria: patients will report average satisfaction as ≥4/5; average appropriateness of the intervention as ≥4/5; ≥75% would recommend FACT to others, and ≥50% indicate they are likely to use FACT strategies following sessions).

Phase 2 To estimate the initial within person change in self-report measures of QOL (QUAL-E), anxiety (GAD-7), depression (CES-D), perceived stress (PSS), perceived social support (ISEL), illness understanding (Prigerson Illness Understanding Scale) and coping strategies (Brief COPE)).

Phase 2 To estimate between group differences in self-report measures of death anxiety (DADDS) and cognitive fusion (CFQ) in patients who participate in FACT intervention compared to a treatment as usual control group. We hypothesize that there will be an initial signal of a group by time effect, where those who participated in FACT report lower scores on DADDS and CFQ compared to those receiving treatment as usual at end-of-treatment and follow-up.

Phase 2 To estimate between group differences in self-report measures of quality of life (QUAL-E), anxiety (GAD-7), depression (CES-D), perceived stress (PSS), perceived social support (ISEL-12), illness understanding (PUQ) and coping strategies (Brief COPE) for those who participated in FACT intervention compared to those receiving treatment as usual.

Exploratory Objectives:

Phase 2 To estimate between group differences in documented goals of care conversations (count) and aggressiveness of medical care within the last 30 days of life for patients after their death with measures defined by the National Quality Forum.

Phase 1 and 2 To estimate between group differences and change over time in concept of double awareness (DAS) and how it may be associated with other self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult cancer patients diagnosed with advanced cancer (solid tumor and hematologic)
* Progressed past at least one line of palliative systemic cancer therapy
* Patient followed by Supportive Care Outpatient Service
* English speaking
* Able to provide written informed consent
* Willing to participate in a stress and coping program
* Willing to identify 1-2 important areas of life they might like to discuss with a counselor
* Moderate levels of death anxiety on DADDS (>=25, on 0-75 scale)
* Access to technology to support institutionally approved video-conferencing platform of Zoom

Exclusion Criteria:

* ECOG performance status >=3 "capable of only limited selfcare; confined to bed or chair more than 50% of waking hours"
* Currently participating in regular psychotherapy (patient defined)
* Documented out of hospital DNR (do not resuscitate) orders
* Presence of active suicidal ideation or need for a higher level of care (as determined by Supportive Care physician or licensed mental health clinician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Kroll, BA,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org